CLINICAL TRIAL: NCT03612505
Title: Caregiver Interventions for Developmental Delays in Young Kenyan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Megan Song McHenry, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1801879405
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Child Development; Parenting; Cognitive Developmental Delay
MeSH Terms: interventions — Child Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Mother groups using principles of UNICEF/World Health Organization's Care for Child Development
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Mother groups using principles of UNICEF/World Health Organization's Care for Child Development — The intervention is expected to occur every two weeks for a total of ten sessions. On the study day, the child- caregiver dyads randomised to intervention group will be shown to the study room. Each intervention session will be estimated to last 90 minutes allocated as follows: 6
  * Introduction (10 minutes)
  * Lesson on *Early Childhood Development* topic (20 minutes)
  * Discussions on strengthens in caregiving around this topic and areas for improvement (30 minutes)
  * Observe caretakers one-on-one in play role with the child (25 minutes)
  * Wrap up/Re-cap (5 minutes) Early Childhood development topics that will be covered include per session are: i) Importance of early childhood development ii) Showing love and building trust iii) Awareness of child's well-being iv) Consistency and daily routines v) Discipline and correction vi) consistency and daily routines vii) Nutrition and cleanliness Viii) Importance of play iX) Dealing with life stresses X) Planning for the future
  Arms: Intervention

SUMMARY:
In this study, the investigators will only administer the intervention to children known to have neurodevelopmental delays. By focusing on adapting the intervention to be only a clinic-based treatment, a small number of community members could be trained to administer the program and increase the potential for sustainability. If the clinic-based group sessions prove to be effective for young children with neurodevelopmental delays, this would help inform the key areas of fidelity needed to maintain effectiveness of the intervention. This study is a critical first step to evaluating the Care for Child Development Intervention (CCDI) program's potential as a cross-cultural intervention that is sustainable and effective for the children at highest risk for neurodevelopmental delay. These results will have significant impacts in improving early childhood neurodevelopment both in Kenya and worldwide.

DETAILED DESCRIPTION:
Objectives:

The broad objective of this proposal is to pilot the CCDI program as an intervention to treat neurodevelopmental delays among 56 young children in Kenya

Specific Aims:

Aim 1: Determine the feasibility of a randomized controlled trial protocol to examine the effectiveness of the CCDI Program for Kenyan children with neurodevelopmental delays aged 18-24 months within a public Maternal-Child Health (MCH) clinic setting.

Hypothesis: The CCDI Program will be feasible, as measured by ≥90% of participants being willing to be randomized to either the intervention or the control group; ≥ 80% attending all 10 biweekly caregiver meetings; ≥80% of children returning for their 6 month follow-up; and ≥80% returning for 12 month follow-up.

Aim 2: Determine the acceptability, facilitators, and barriers of the CCDI Program for use in eligible children.

Hypothesis: The CCDI Program will be acceptable, as determined by an analysis of prospective, concurrent, and retrospective acceptability, and specific facilitators and barriers to the program will be identified. Using focus group discussions and semi-structured interviews with caregivers, clinical providers, and community leaders, the investigators will determine aspects of the program are acceptable, facilitators, and barriers to improved neurodevelopmental care and allow the CCDI program to function optimally in this setting.

Aim 3: Estimate the effect size of the CCDI Program to reduce neurodevelopmental delays in young Kenyan children.

Hypothesis: The investigators will demonstrate a 40% decrease in the number of children with neurodevelopmental delays, as determined by a culturally adapted Bayley Scales of Infant and Toddler Development, 3rd edition (BSID-III) standardized score with implementation of the CCDI Program. This data will inform sample size justification for a future intervention study.

ELIGIBILITY:
Inclusion Criteria:

* age 18-24 months
* communicate in either English or Kiswahili
* Score < 85 on one of the BSID-III subscales (mild/moderate/severe delay in cognitive, motor, or language).
* Have a caregiver who can communicate in English or Kiswahili
* Have a caregiver responsible for child's daily activities

Exclusion Criteria:

* Profound neurological impairment, such as severe cerebral palsy, deafness, or blindness preventing them from participating in the groups.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Bayley Scales of Infant and Toddler Development, 3rd edition (BSID-III) scores | Baseline, 6 months, 12 months
  Measures cognitive, language, and motor development. Composite scores for cognitive (range of scores 55-145), language (range of scores 47-153), and motor (range of scores 46-154) development. Lower scores indicate worse development. Subscales (e.g. fine and gross motor for motor and expressive and receptive language for language) are summed to create the composite score.

SECONDARY OUTCOMES:
Change In Perspectives around Child Development, gathered by Focus Group Discussions | Baseline and 6 months
  Qualitative interviews with caregivers in Group 1, who will receive the intervention during the first 6 months of the study. Qualitative interviews will also be performed with Group 2 to see if there were any changes in perspectives on child development without the intervention
Change In Perspectives around Child Development, gathered by Focus Group Discussions | 6 months and 12 months
  Qualitative interviews with caregivers in Group 2, who will receive the intervention during the second 6 months of the study. Qualitative interviews will also be performed with Group 1 to see if there were any changes in perspectives on child development after the intervention has ceased
Change in mother interactions, gathered by video-taped mother interactions | Baseline and 6 months
  Coding of mother's interactions with children while waiting. We will compare Group 1, who will receive the intervention during the first 6 months, as well as Group 2, who will not be receiving the intervention during this interval
Change in mother interactions, gathered by video-taped mother interactions | 6 months and 12 months
  Coding of mother's interactions with children while waiting. We will compare Group 2, who will receive the intervention during the first 6 months, as well as Group 1, who had received the intervention but not longer is receiving it in the second 6 months.
Change in Home Observations Measurement of the Environment (HOME) scores | Baseline, 6 months, 12 months
  Structured observations and questions performed in a families home. Subscales are as follows: Responsivity (score range 0-11), acceptance (0-8), organization (0-6), learning materials (0-9), involvement (0-6), variety (0-5). The lower scores indicate worse performance. These subscales are summed to give the total score.
Change in MacArthur-Bates Communication Developmental Inventory (CDI) scores | Baseline, 6 months, 12 months
  Language. Scale range is 0-100, with the lower scores indicating worse performance. No subscales will be used in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University School of Medicine, Eldoret, Uasin Gishu County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
I'm happy to share the data but I'm not sure of the best means of doing this